CLINICAL TRIAL: NCT07283874
Title: Does it Matter the Volume of Injectate on the Outcome of Ultrasound-guided Perineural Injection for Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Kamal Abdullah Mohamed, Resident doctor at Anesthesia, Intensive Care and Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: volume of injectate CTS
Record Dates: First submitted 2025-12-07; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): wrists undergoing ultrasound guided perineural injection of 5 ml total volume of injectate (3ml dextrose 5% +1 ml Triamcinolone acetonide + 1 ml lidocaine 2%) for carpel tunnel syndrome
  Interventions: Drug: Dextrose 5%; Drug: Triamcinolone Acetonide (Aristocort® C); Drug: Lidocaine 2 %
- Group B (Active Comparator): wrists undergoing ultrasound guided perineural injection of 10 ml total volume of injectate (8 ml dextrose 5% +1 ml Triamcinolone acetonide + 1 ml lidocaine 2%) for carpel tunnel syndrome
  Interventions: Drug: Dextrose 5%; Drug: Triamcinolone Acetonide (Aristocort® C); Drug: Lidocaine 2 %

INTERVENTIONS:
Drug: Dextrose 5% — patients injected with 8ml dextrose 5%
  Arms: Group A
Drug: Dextrose 5% — patients injected with 3 ml dextrose 5%
  Arms: Group B
Drug: Triamcinolone Acetonide (Aristocort® C) — patients injected with 1 ml Triamcinolone acetonide
Drug: Lidocaine 2 % — patients injected with 1ml lidocaine 2%)

SUMMARY:
Carpal tunnel syndrome (CTS) is an entrapment neuropathy affecting the median nerve with a lifetime prevalence of about 8% in the adult population. Carpal tunnel syndrome (CTS) occurs with the symptoms of intermittent nocturnal paresthesia and dysesthesia, followed by loss of sensation, weakness, and thenar muscle atrophy in later stages.

Although the etiology of CTS is multifactorial, compression of the median nerve in a space-limited osteofibrous canal at wrist level was proposed.

The gold standard of diagnosis is electrophysiological study, but ultrasonography was applied in recent decades for a better approach to the morphology change of the median nerve.Nerve hydrodissection (HD) is a widely used technique that involves the injection of fluid to separate the nerve from the surrounding structures.

HD is now considered a novel approach for the treatment of CTS with safe and outstanding long-term effects. A potential benefit of HD is to release the pressure on the "free nerves supplying the main nerves," called "nervi nervorum." Early, the compression of the vasa nervorum would affect venous outflow, causing the accumulation of toxins in the affected part. Then, the lymphatic drainage, located outside the epineurium, would undergo compressive effects.

HD can also decrease the gliding resistance of the median nerve within the carpal tunnel, which is considered a principal patho-mechanical cause of nerve injury.

Hydrodissection HD of the entrapped median nerve is considered a safe and efficacious approach for treatment of mild to moderate CTS and could be offered to patients with severe CTS if surgery is refused or can't be done due to other medical comorbidities. The use of US-guided HD could improve symptom severity, functional status, and the US parameters of nerve entrapment. HD has a long-term efficacy outcome; 88.6% of patients reported an effective outcome, and this may vary according to the initial severity status.

Different types of injectants are available and studied, with no clear indication of use for each type. However, PRP, D5W, and HA were more efficient than NS as regards subjective and objective improvement. PRP and HA were more effective for long-term nerve recovery, while HA was preferred for the earliest response. So, we recommend making the choice based on every patient's severity scale and electrophysiological scales, which means that for patients with mild forms and severe pain.

Injection of a large volume could be a better option in order to dissect a larger area, provide a better environment for the nerve repair mechanisms, and release the vascular and neural compressive elements.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-80 years old 2. Patients diagnosed with idiopathic CTS. 3. Abnormal electrophysiological analysis showing mild to moderate CTS 4. Symptoms and signs including:

  1. pain or paraesthesia in the median nerve innervated area (at least two digits with such symptoms between the thumb and the 4th digit) for more than 6 months not responding to conservative management including (vitamin B complex, nonsteroidal anti-inflammatory drugs, oral steroids, and/or night splint)
  2. positive Phalen test, Tinel sign, or flick sign
  3. The patient's initial examination was based on the American Academy of Orthopaedic Surgeons Clinical Practice Guideline recommendations prior to their inclusion and confirmed by nerve conduction studies

Exclusion Criteria:

* 1- Age less than 20 years 2- severe CTS (abductor policies brevis muscle atrophy with distal latency time >6.5 MS).

  3- MN electrophysiology study revealing absent potentials. 4- its cross-sectional area (CSA) >15 mm2 by sonographic checkup. 5- previous surgery of carpal tunnel. 6- previous wrist injection within 3 months 7- history of peripheral nerve injuries (brachial plexopathy, cervical radiculopathy or thoracic outlet syndrome) 8- CTS due to systemic causes, for example, endocrinal and/or pregnancy, rheumatoid arthritis, gouty or psoriatic osteoarthritis.

  9- concurrent use of antihistaminic, or cortisone. 10- Participant refusal. 11- local infection. presence of coagulopathy, and/or allergy to the included medications were also points for patients' exclusion from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the severity of pain in patients with Carpal Tunnel Syndrome | 1 month
  Pain assessment through the VAS was explained to the patient (through selection of the number that represents his/her pain with 0 = no pain, and 10 = worst pain